CLINICAL TRIAL: NCT07077993
Title: The Relationship Between Lower Extremity Strength, Dynamic Balance, and Core Endurance in Elite Youth Rowers: A Cross-Sectional Observational Study
Brief Title: "Muscle Strength, Balance, and Core Endurance in Elite Adolescent Rowers: A Cross-Sectional Study"
Acronym: REBCORE
Status: Completed | Type: Observational
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Burçin Uğur Tosun, Principal Investigator PhD Physiotherapist Burcin Ugur Tosun, Eastern Mediterranean University
Other Study IDs: 2025-06
Record Dates: First submitted 2025-07-12; First posted 2025-07-22 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Neuromuscular Function; Postural Balance; Core Stability; Muscle Strength
Keywords: Rowing Performance; Core Endurance; Dynamic Balance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Male Athletes: Elite male adolescent rowers (n=36), aged 16-18, participating in national-level rowing training at least 5 times per week.
- Female Athletes: Elite female adolescent rowers (n=32), aged 16-18, participating in national-level rowing training at least 5 times per week.

SUMMARY:
This study aims to investigate the relationship between lower extremity isokinetic strength, dynamic balance, and core muscle endurance in elite adolescent rowers aged 14-17. A total of 68 athletes (31 males, 37 females) will be assessed through standardized protocols involving isokinetic testing, the Y Balance Test, and McGill Core Endurance Tests. The study aims to contribute to performance monitoring and injury prevention strategies in rowing sports.

DETAILED DESCRIPTION:
This observational cross-sectional study aims to investigate the relationships between lower extremity muscle strength, dynamic balance, and core endurance in elite adolescent rowers aged 14-17. A total of 68 rowers (32 females, 36 males) licensed by the Turkish Rowing Federation were included. All participants had a minimum of two years of rowing experience and trained at least four days per week.

Lower extremity muscle strength was assessed using isokinetic dynamometry at angular velocities of 60°/s and 300°/s. Core endurance was evaluated using the McGill Core Endurance Test Battery, including trunk flexor, extensor, and lateral plank tests. Dynamic balance was assessed via the Y Balance Test and normalized to leg length.

The study also examined potential sex-based differences in neuromuscular performance and investigated inter-variable correlations among muscle strength, balance, and core endurance. In addition, asymmetry in dynamic balance performance was analyzed as a risk factor for performance and injury.

This study is expected to provide practical insights for sports physiotherapists and coaches working with adolescent rowers, particularly in optimizing performance and designing sex-specific injury prevention strategies.

ELIGIBILITY:
Inclusion Criteria:

Elite adolescent rowers aged 16 to 18 years

Licensed athletes training at least 5 days per week

Registered with a national-level rowing team or rowing education program

Minimum 2 years of regular rowing experience

No current musculoskeletal or neurological injury

Voluntary participation with informed consent (parental consent required for minors)

Exclusion Criteria:

History of lower extremity or spinal surgery

Current injury or condition affecting strength, balance, or posture

Diagnosed neurological disorder or vestibular dysfunction

Acute illness, severe fatigue, or muscle soreness on the day of testing

Active menstruation phase in female participants on the day of testing

Lack of cooperation or unwillingness to follow instructions

Ages: 16 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — This study includes both male and female elite adolescent rowers aged 16-18. A gender-based comparative analysis was planned to examine potential sex-specific differences in muscle strength, core endurance, and dynamic balance performance. Both sexes were evaluated separately to identify neuromuscular characteristics and training needs unique to each group.
Study Population: The study population consists of 68 elite adolescent rowers (32 females, 36 males) aged 16 to 18 years, actively competing and training under the Turkish Rowing Federation. All participants were healthy, licensed athletes with at least two years of regular rowing experience and were training at least five times per week at a national-level rowing training center.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-07-20 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Composite Y Balance Test Score (%) | Cross-sectional assessment at baseline (single visit)
  Dynamic balance will be assessed using the Y Balance Test. Reach distances in three directions will be normalized to limb length, and a composite balance score will be calculated. The outcome will be used to compare balance performance across sex groups.
Isokinetic Quadriceps Peak Torque at 60°/s (Nm) | Cross-sectional assessment at baseline (single visit)
  Peak torque of the dominant quadriceps muscle will be measured using an isokinetic dynamometer at an angular velocity of 60°/s. The outcome will be recorded in Newton-meters (Nm) and used to analyze muscle strength differences between groups.
Core Extensor Endurance Time (seconds) | Cross-sectional assessment at baseline (single visit)
  Trunk extensor endurance will be evaluated using the McGill Trunk Extensor Endurance Test. Participants will maintain a horizontal prone posture over the edge of a bench with the pelvis stabilized. The maximum time (in seconds) that the position can be held with proper form will be recorded as the endurance score.

CONTACTS AND LOCATIONS:
Overall Officials: burcin ugur tosun, PHD, Principal Investigator — Ministry of Youth and Sports, Olympic Preparation Center, Adana, Türkiye; gulhan yilmaz gokmen, Assoc. Prof, Study Chair — Faculty of Health Sciences, Bandırma Onyedi Eylül University, Bandırma, Balıkesir, Türkiye
Locations (1):
- Burcin Ugur Tosun, Famagusta, Cyprus